CLINICAL TRIAL: NCT06786468
Title: Randomized Controlled Trial of Standard Care With or Without Early Palliative Care Provided by Palliative Care Specialist in Advanced Non-small Cell Lung Cancer Patients
Brief Title: Standard Care With or Without Early Palliative Care Provided by Palliative Care Specialist in Advanced Non-small Cell Lung Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 068/2567(IRB3)
Record Dates: First submitted 2025-01-06; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer - Non Small Cell; Lung Cancer (NSCLC)
Keywords: early palliative care; palliative care; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early palliative care with standard care (Experimental): The patients will attend palliative care clinic once a month during the first three months together with oncology clinic visits
  Interventions: Other: Early palliative care integration; Drug: Standard systemic treatment for advanced lung cancer
- Standard care (Active Comparator): The patients will attend oncology clinic as usual
  Interventions: Drug: Standard systemic treatment for advanced lung cancer

INTERVENTIONS:
Other: Early palliative care integration — The patients will attend palliative care clinic once a month during the first three months together with routine oncology clinic visits
  Arms: Early palliative care with standard care
Drug: Standard systemic treatment for advanced lung cancer — Standard systemic treatment for advanced lung cancer

SUMMARY:
Early palliative care has been shown to improve the survival of advanced lung cancer patients. However, most of the clinical studies were performed in the era when systemic treatment options for this disease were limited. Currently, many effective treatment options are available, including targeted therapy and immunotherapy. These novel agents improve the treatment outcomes while having less toxicity compared to conventional chemotherapy. Moreover, medical oncologists are now trained to provide palliative care for patients. This study was designed to demonstrate whether early palliative care provided by the palliative care specialist still improves the quality of life or survival of advanced lung cancer patients compared to standard care provided by the medical oncologist.

DETAILED DESCRIPTION:
Advanced non-small cell lung cancer patients initiating a systemic treatment will be randomized to the early palliative care arm (attending a palliative care clinic once a month during the first three months concurrently with oncology clinic appointment) or the standard care arm (attending oncology clinic only). The patients will be asked to complete the quality of life questionnaires (FACT-L, EQ-5D-5L), mental health questionnaire (PHQ-9), and pain assessment once a month for three months and at the sixth month.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years old
* Pathologically confirmed advanced non-small cell lung cancer
* Plan to receive systemic treatment for lung cancer within three weeks
* ECOG performance status 0-2 with estimated life expectancy > 24 weeks
* Having at least 4 scores according to Edmonton Symptom Assessment System (ESAS)
* Able to complete the questionnaires

Exclusion Criteria:

* Had received systemic treatment for advanced lung cancer before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Quality of life score (FACT-L Total Score) | 12 weeks after treatment
  The patients were asked to assess their Health-related Quality Of Life (HRQoL) using FACT-L (Functional Assessment of Cancer Therapy - Lung) questionnaire. The score ranges from 0-136 with higher score indicating better HRQoL.

SECONDARY OUTCOMES:
Change in quality of life (FACT-L Total Scores) | 12 and 24 weeks after treatment
  The patients were asked to assess their Health-related Quality Of Life (HRQoL) using FACT-L (Functional Assessment of Cancer Therapy - Lung) questionnaire. The score ranges from 0-136 with higher score indicating better HRQoL. Change in FACT-L Total Scores defined as the difference between FACT-L Total Score at a specified time point minus baseline FACT-L Total Score.
Change in mental health score (PHQ-9) | 12 and 24 weeks after treatment
  The patients were asked to assess their depression levels using a Patient Health Questionnaire 9 (PHQ-9). The score ranges from 0-27 with 0 indicating no depression and 27 indicating severe depression.
Change in pain score | 12 and 24 weeks after treatment
  The patients were asked to assess their pain using a Numerical Rating Scale (NRS). The score ranges from 0-10 with 0 indicating no pain and 10 indicating worst pain imaginable.
One-year survival rate | One year after treatment
Two-year survival rate | Two years after treatment
Proportion of patients who have advanced care plan | six months
Change in utility score measured by EQ-5D-5L questionnaire | 12 and 24 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lucksamon Thamlikitkul, MD, PhD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No